CLINICAL TRIAL: NCT05173285
Title: Feasibility and Acceptability of a Brief Internet-Based Acceptance and Commitment Therapy Intervention for Parents in the Postpartum: A Feasibility Randomized Control Trial
Brief Title: Brief Internet-Based Acceptance and Commitment Therapy Intervention for Parents in the Postpartum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannah Palma Carlos (Other)
Responsible Party: Sponsor-Investigator, Hannah Palma Carlos, Principal Investigator, Royal Holloway University
Organization: Royal Holloway University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 27112020
Record Dates: First submitted 2021-11-05; First posted 2021-12-29 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Online ACT Intervention (Experimental): Intervention Condition: Participants in this arm will take part in a brief ACT intervention delivered online via Qualtrics across 4-weeks; one session per week. The first two weeks will focus on mindfulness, with participants being invited to practice formal (i.e. 3-minute breathing exercise) and informal mindfulness practices (e.g. mindful walking, mindful drink etc.) during the week. The final two weeks will focus on values, specifically supporting participants to identify their personal values and set goals relating to these values. Participants have up to 6 weeks to complete the 4-week intervention.
  Interventions: Diagnostic Test: Baseline Assessment; Behavioral: Brief Online ACT Intervention; Diagnostic Test: Post-Intervention Assessment (i.e. between 4-6 weeks after baseline assessment); Diagnostic Test: Follow-up Assessment (i.e. between 8-12 weeks after baseline assessment)
- Waitlist Control (Other): Control Condition: Participants in this arm will not receive an intervention. They will however, been given access to the brief online ACT intervention at the end of study.
  Interventions: Diagnostic Test: Baseline Assessment; Diagnostic Test: Post-Intervention Assessment (i.e. between 4-6 weeks after baseline assessment); Diagnostic Test: Follow-up Assessment (i.e. between 8-12 weeks after baseline assessment)

INTERVENTIONS:
Diagnostic Test: Baseline Assessment — At baseline (i.e. Pre-intervention) participants will complete several questionnaires online via Qualtrics.
Behavioral: Brief Online ACT Intervention — Participants will complete the 4-week online intervention via Qualtrics
  Arms: Brief Online ACT Intervention
Diagnostic Test: Post-Intervention Assessment (i.e. between 4-6 weeks after baseline assessment) — Participants will complete several questionnaires online via Qualtrics.
Diagnostic Test: Follow-up Assessment (i.e. between 8-12 weeks after baseline assessment) — Participants will complete several questionnaires online via Qualtrics.

SUMMARY:
It is common for parents in the postpartum period (the first twelve months following childbirth) to experience psychological difficulties, particularly low mood. Acceptance and Commitment Therapy (ACT) is an evidence-based intervention that aims to cultivate psychological flexibility; the ability to stay in contact with the present moment regardless of unpleasant thoughts, feelings and bodily sensations, while choosing one's behaviours based on values. Acceptance and Commitment Therapy (ACT) is effective in reducing depression in the general population, including brief ACT interventions. However, the effectiveness of ACT interventions in the postpartum period is not yet fully established.

This study aims to investigate the feasibility (recruitment source, rate and attrition rate), acceptability (usability, usefulness and satisfaction) and the potential effectiveness (to inform the required sample size for a fully powered randomised control trial) of a four week internet-based ACT intervention for postpartum parents on depression.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Have a child under 12 months
* Scoring 10 or above on the Edinburgh Postnatal Depression Scale
* Access to the internet through a computer, tablet or phone
* Fluency in English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Change in Depression on The Edinburgh Postnatal Depression Scale from Baseline to Post Intervention (i.e. between week 4-6 after baseline assessment) | Baseline and Between 4 to 6 Weeks
  The Edinburgh Postnatal Depression Scale is a 10-question self-rating questionnaire measuring severity of postpartum depression symptoms. Change = (Between 4 to 6 Weeks- Baseline Score)
Change in Depression on The Edinburgh Postnatal Depression Scale from Baseline to Follow-up (i.e. between week 8-12 after baseline assessment) | Baseline and Between 8 to 12 Weeks
  The Edinburgh Postnatal Depression Scale is a 10-question self-rating questionnaire measuring severity of postpartum depression symptoms. Change = (Between 8 to 12 Weeks- Baseline Score)

SECONDARY OUTCOMES:
Change in Wellbeing Score on The Flourishing Scale from Baseline to Post Intervention (i.e. between week 4-6 after baseline assessment) | Baseline and Between 4 to 6 Weeks
  The Flourishing scale provides a single psychological well-being score. Participants answer on a 7-point scale to what extent they agree (7) or disagree (1) with the 8 statements relating to relationships, self-esteem, purpose and optimism. Change = (Between week 4 to 6- Baseline Score)
Change in Wellbeing Score on The Flourishing Scale from Baseline to Follow Up (i.e. between week 8-12 weeks after baseline assessment) | Baseline and Between 8 to 12 Weeks
  The Flourishing scale provides a single psychological well-being score. Participants answer on a 7-point scale to what extent they agree (7) or disagree (1) with the 8 statements relating to relationships, self-esteem, purpose and optimism. Change = (Between week 8 to 12- Baseline Score)

OTHER OUTCOMES:
Change in Mindfulness skills on The Five Facet Mindfulness Questionnaire from Baseline to Post Intervention (i.e. between week 4-6 after baseline assessment) | Baseline and Between 4 to 6 Weeks
  39-item questionnaire measures describing, non-reactivity, act with awareness, non-judging and observing. Items are rated on a 5-point scale ('1' -never or very rarely true, '5'- very often or always true). This study will include 31 items from the questionnaire, as it will not include the Observer factor items. This measure will be used to explore intervention specific changes in mindfulness skills.
  Change = (Between week 4 to 6- Baseline Score)
Change in Mindfulness skills on The Five Facet Mindfulness Questionnaire from Baseline to Follow Up (i.e. between week 8-12 after baseline assessment) | Baseline and Between 8 to 12 Weeks
  39-item questionnaire measures describing, non-reactivity, act with awareness, non-judging and observing. Items are rated on a 5-point scale ('1' -never or very rarely true, '5'- very often or always true). This study will include 31 items from the questionnaire, as it will not include the Observer factor items. This measure will be used to explore intervention specific changes in mindfulness skills.
  Change = (Between Week 8 to 12- Baseline Score)
Change in Valued Living on The Valuing Questionnaire from Baseline to Post Intervention (i.e. between week 4-6 after baseline assessment) | Baseline and Between 4 to 6 Weeks
  The Valuing Questionnaire is a 10-item questionnaire measuring personal values enactment during the past week. The Valuing Questionnaire measures two constructs; progress in valued living and obstruction to valued living.
  Change = (Between Week 4 to 6 - Baseline score)
Change in Valued Living on The Valuing Questionnaire from Baseline to Follow Up (i.e. between week 8-12 after baseline assessment) | Baseline and Between 8 to 12 Weeks
  The Valuing Questionnaire is a 10-item questionnaire measuring personal values enactment during the past week. The Valuing Questionnaire measures two constructs; progress in valued living and obstruction to valued living.
  Change = (Between Week 8 to 12 - Baseline score)
System Usability Scale (SUS) System Usability Scale (SUS) System Usability Scale | Between 4 to 6 Weeks from Baseline Assessment
  This 10-item questionnaire asks participants to rate on a 5-point Likert Scale positive and negative descriptions of the intervention.
Usefulness of the online intervention | Between 4 to 6 Weeks from Baseline Assessment
  Participants asked to rate usefulness (i.e. "I found this intervention useful") on a 5-point Likert scale (1= strongly disagree - 5= strongly agree).
Satisfaction with the online intervention | Between 4 to 6 Weeks from Baseline Assessment
  Participants asked to select all applicable items from a list of items relating to ways the intervention met or failed their expectations.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Palma Carlos, Principal Investigator — Royal Holloway University
Locations (1):
- Royal Holloway University of London, Egham, Surrey, United Kingdom